CLINICAL TRIAL: NCT05723328
Title: The Effect of a Group Music Therapy Advocacy Recording Intervention (MTAR) on Internalized Stigma in Adult Psychiatric Inpatients in Acute Care
Brief Title: Music Therapy Advocacy Recording Intervention (MTAR) on Internalized Stigma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Resource Limitations
Sponsor: Hackensack Meridian Health (Other)
Collaborators: American Music Therapy Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro2022-0570
Record Dates: First submitted 2023-02-01; First posted 2023-02-10 (Actual); Results first posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: Mental Health Issues; Bipolar Disorder; Depressive; Schizophrenia Spectrum and Other Psychotic Disorders; Anxiety Disorder
Keywords: Internalized stigma; Music therapy; Music Therapy Advocacy Recording Intervention; Schizophrenia Spectrum and Other Psychotic Disorders; Mental Health Issues
MeSH Terms: conditions — Bipolar Disorder; Schizophrenia Spectrum and Other Psychotic Disorders; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Pseudo cluster randomized controlled design (Borm et al., 2005) will take advantage of the unit's two separate residential areas
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): The intervention consists of a sequence of five music therapy song-writing and recording groups, one per day. Internalized stigma will be assessed within 3 days of admission (pretest/baseline), at ten days (posttest), and at 3 weeks from baseline (follow-up), using the Internalized Stigma of Mental Illness Inventory.
  Interventions: Behavioral: Group Music Therapy Advocacy Recording Intervention (MTAR)
- Control Group (No Intervention): Access to standard of care services that include several groups per day focused on topics of coping skills, mindfulness, journaling, creative arts, wellness recovery, recreation, and at least one music therapy group.

INTERVENTIONS:
Behavioral: Group Music Therapy Advocacy Recording Intervention (MTAR) — Music Therapy Advocacy Recording Intervention (MTAR) is a sequence of group music therapy song-writing and recording sessions framed as a mental health awareness project to be shared with the general public.
  Arms: Treatment Group

SUMMARY:
This study will use a systematic music therapy intervention on patients with mental illness trying to help them with their internalized stigma.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the effect of a systematic music therapy intervention on internalized stigma of mental illness. The secondary objective is to evaluate the potential for the treatment effect to vary across subject diagnostic categories. This study will also examine the ability of the treatment effect to persist after 3 weeks as an exploratory objective.

Data collection will be conducted in the Acute Care Unit (ACU) of Hackensack Meridian Health Carrier Clinic (HMHCC) over a period of ten months. Subjects will be drawn from the pool of patients admitted to the HMHCC ACU during that time. Adults aged 18-65 with severe mental illness with a diagnosis of bipolar or a related disorder, depressive or anxiety disorder, or schizophrenia spectrum or other psychotic disorders as defined by the Diagnostic and Statistical Manual of Mental Disorders version 5 (DSM-5 : 5th ed.; American Psychiatric Association, 2013), of prolonged duration with a significant degree of disability or social dysfunction (Ruggeri et al., 2000) are eligible to participate. Eligible participants must be able to provide informed consent as determined by the doctor.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the HMHCC ACU
* Able to read and comprehend the ISMI questionnaire, provide informed consent,
* With a severe mental illness of prolonged duration with a significant degree of disability or social dysfunction

Exclusion Criteria:

* Patients on S1 status (1:1 patient observation) or isolation protocol
* Evidence of organic brain disease, severe acute symptomatology, hearing deficit, and intellectual disability.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zachary D Fischer, PhD, MT-BC, Principal Investigator — Hackensack Meridian Health
Locations (1):
- Carrier Clinic, Belle Mead, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Consented Patients Randomized to Unit W: Patients consented for the Music Therapy Advocacy Recording Intervention (MTAR) on Internalized Stigma randomized to ACU West
- Consented Patients Randomized to Unit E: Patients consented for the Music Therapy Advocacy Recording Intervention (MTAR) on Internalized Stigma randomized to ACU East
Period: Overall Study
Arm/Group | Consented Patients Randomized to Unit W | Consented Patients Randomized to Unit E
Started | 5 | 2
Received Music Therapy | 0 | 0
Completed | 0 | 0
Not Completed | 5 | 2
Not completed — Investigator's Decision | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Consented Patients: Patients consented for the Music Therapy Advocacy Recording Intervention (MTAR) on Internalized Stigma by not randomized
Arm/Group | Consented Patients
Number analyzed (Participants) | 7
Age, Customized [Median (Full Range); unit: years] | 40 [26 to 64]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
  Non-binary | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in the Internalized Stigma of Mental Illness Inventory (ISMI) Score Between Pre and Post MTAR
Description: The Internalized Stigma of Mental Illness Inventory will be administered before and after the MTAR intervention and the change in the score will be reported.
  Primary outcome will be reported only for the treatment arm. The internalized stigma of mental illness inventory is a 29 item questionnaire. Items are scored on a 1-4 scale, with the total scale score calculated as a sum of the items then dividing by the total number of answered items.
Time Frame: Post MTAR intervention (day 8-10)
Population: Study interventions never took place
Arm/Group | Consented Patients
Number analyzed (Participants) | 0

2. Secondary Outcome: Change in the ISMI Score Based on Diagnostic Category
Description: Change in the Internalized Stigma of Mental Illness Inventory (ISMI) score between pre and post MTAR across subject diagnostic categories. ISMI scores will be compared between subjects with no diagnosis or diagnosed with schizophrenia spectrum and other psychotic disorders, bipolar and related disorders, depressive disorders, and anxiety disorders, as classified by the American Psychiatric Association's Diagnostic and Statistical Manual of Mental Disorders - 5th edition (DSM-5; American Psychiatric Association, 2013).
  The internalized stigma of mental illness inventory is a 29 item questionnaire. Items are scored on a 1-4 scale, with the total scale score calculated as a sum of the items then dividing by the total number of answered items.
Time Frame: Post MTAR intervention (day 8-10)
Population: Study procedures never took place
Arm/Group | Consented Patients
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 10 days post admission
Description: No study procedures were initiated and no music therapy intervention was introduced to study participants.
Groups:
- Consented Patients: Patients consented but not received the the Music Therapy Advocacy Recording Intervention (MTAR) on Internalized Stigma
Arm/Group | Consented Patients
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-20): https://cdn.clinicaltrials.gov/large-docs/28/NCT05723328/Prot_SAP_000.pdf